CLINICAL TRIAL: NCT03675867
Title: Exercise and Baseline Respiratory Functional Tests Among Obese Teenagers
Acronym: EFRADO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2018/390
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese teenagers
  Interventions: Other: Correlation between resting respiratory parameters and cardio-respiratory parameters at exercise

INTERVENTIONS:
Other: Correlation between resting respiratory parameters and cardio-respiratory parameters at exercise — Correlation between resting respiratory parameters and cardio-respiratory parameters at exercise

SUMMARY:
In obese adolescents, the severity of obesity should not influence the outcome of resting PFT. The amplitudes of the rest PFT should make it possible to predict the performance achieved while exercising on a cycloergometer.

We wish to highlight the presence of a significant correlation, probably low, between some respiratory parameters at rest, and cardio-vascular parameters at the exercise.

ELIGIBILITY:
Inclusion Criteria:

* Children aged >12 y.o and <18 y.o
* BMI > 30
* with a previous pulmonary function test (PFT) available in the medical record

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Obese teenagers with previous PFT available in the medical record
Sampling Method: Non-Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2018-08-16 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Correlation between resting respiratory parameters and cardio-respiratory parameters at exercise | Day 1
  Correlation between resting respiratory parameters: total lung capacity (TLC), forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and cardio-respiratory parameters at exercise: maximal oxygen uptake (VO2 max), power achieved during incremental testing (Pmax), blood gas, at the time of the pulmonary function test.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Degano, MD PhD, Principal Investigator — CHU de Besançon
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No